CLINICAL TRIAL: NCT02450084
Title: Postoperative Analgesic Effects of Ultrasound-guided Bilateral Rectus Sheath Block for Robotic Single-port Gynecologic Surgery
Brief Title: Ultrasound-guided Bilateral Rectus Sheath Block for Robotic Single-port Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Youn Jin Kim, Associate Professor of Anesthesiology and Pain Medicine, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EUMC 2015-01-024-002
Record Dates: First submitted 2015-05-08; First posted 2015-05-21 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female | interventions — Ropivacaine; Bandages

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rectus sheath block (Experimental): Patients of RSB group will be performed ultrasound-guided bilateral RSB after induction of general anesthesia. After draping the needle insertion site, a 22-gauge, 50-mm needle will be inserted medial to the probe by the in-plane technique and advanced in a lateral direction on just lateral to umbilicus. 15 ml of 0.25% ropivacaine will be injected on the posterior border of rectus muscle. This procedure will be performed bilaterally and total 30 ml of 0.25% ropivacaine will be injected. After the surgery, a bandage will be attached on injection site where is same as the incision site of surgery. All patients will use total 100 ml of IV-PCA containing fentanyl 800 µg for 48 hours postoperatively.
  Interventions: Procedure: Rectus sheath block; Drug: Ropivacaine; Other: Bandage; Drug: IV-PCA containing Fentanyl
- Control (Sham Comparator): Patients of Control group will be proceeded a surgery scheduled after induction of general anesthesia without any procedure such as placebo injection. After the surgery, a bandage will be attached on the incision site where is same as the block injection site of RSB group. All patients will use total 100 ml of IV-PCA containing fentanyl 800µg for 48 hours postoperatively.
  Interventions: Other: Bandage; Drug: IV-PCA containing Fentanyl

INTERVENTIONS:
Procedure: Rectus sheath block — Ultrasound-guided bilateral rectus sheath block of RSB group using 0.25% Ropivacaine
  Other Names: RSB
  Arms: Rectus sheath block
Drug: Ropivacaine — Ultrasound-guided bilateral rectus sheath block of RSB group using 0.25% Ropivacaine
  Other Names: Naropin
  Arms: Rectus sheath block
Other: Bandage — After the surgery, a bandage will be attached on injection site where is same as the incision site of surgery.
Drug: IV-PCA containing Fentanyl — All patients will use total 100 ml of IV-PCA containing 800 µg of fentanyl for 48 hours postoperatively.
  Other Names: Intravenous patient controlled analgesia using fentanyl

SUMMARY:
Rectus sheath block (RSB) is a kind of anterior abdominal wall block. It has postoperative analgesic effect for abdominal surgery with midline incision. Robotic gynecologic surgery is accompanied by significant postoperative pain and usually IV-PCA is used to manage the pain.The purpose of this study is to investigate the analgesic effect of ultrasound-guided RSB to single-port robotic gynecologic surgery which has incision site at umbilical area. Patients will randomly assigned to two groups, RSB group and Control group. Each patients will assessed for time to first rescue analgesia, verbal numerical rating pain scores, number of rescue analgesic demands, and postoperatively opioids use by IV-PCA by a blinded investigator at 0, 1, 6, 12, 24 and 48 hours postoperatively.

DETAILED DESCRIPTION:
Patients of RSB group will be performed ultrasound-guided bilateral RSB after induction of general anesthesia. The procedure will be performed bilaterally and 15 ml on each side, total 30 ml of 0.25% ropivacaine will be injected. After the procedure, a surgery scheduled will be proceeded. Patient of Control group will be proceeded the surgery after induction of anesthesia. All patients will use total 100 ml of IV-PCA containing 800 µg of fentanyl for 48 hours postoperatively. If a patient complains pain more intense than VNRS 4 or demands an analgesic drug, a rescue analgesic would be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Robotic single-port gynecologic surgery
* American society of Anesthesiologists (ASA) physical status classification I-II
* Age: 21-60

Exclusion Criteria:

* Gynecologic cancer operation
* History of previous abdominal surgery
* Allergy to local anesthetics(ropivacaine)
* Opioid tolerance
* Coagulopathy
* Infection at the needle insertion site
* Difficulty to cooperating

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Verbal numerical rating scale | 6 hours postoperatively
  Postoperative pain on each time point which is expressed by verbal numerical rating scale (0 ~ 10)

SECONDARY OUTCOMES:
Total opioids use | 0, 1, 6, 12, 24, 48 hours postoperatively
  Total dosage of injected fentanyl through IV-PCA
Time to first rescue analgesic request | 48 hours postoperatively
  How long it takes postoperative time to first additional analgesic drug injection by patient's request
Verbal numerical rating scale | 0, 1, 12, 24, 48 hours postoperatively
  Postoperative pain on each time point which is expressed by verbal numerical rating scale (0 ~ 10)

CONTACTS AND LOCATIONS:
Overall Officials: Youn Jin Kim, MD, PhD, Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea